CLINICAL TRIAL: NCT07192965
Title: ECG-less Coronary Computed Tomography Angiography in the Management of Patients Presenting With High-troponin Chest Pain
Acronym: ECLECTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Francesco Giangiacomi, Medical Doctor, fellow in interventional cardiology, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1432025000119
Record Dates: First submitted 2025-09-13; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Chest Pain; Acute Coronary Syndromes (ACS)
Keywords: Chest pain; Acute coronary syndrome; NSTEMI; ECG-less coronary computed tomography angiography; ECG-les CCTA
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm (Other): All patients will be before scanned with a ECG-less CCTA and then undergo invasive coronary angiography. There is one single arm.
  Interventions: Radiation: Non-ECG-gated computed tomography

INTERVENTIONS:
Radiation: Non-ECG-gated computed tomography — Scanning with a Revolution Apex Elite system (GE Healthcare, WI, USA), using hyperdrive pulmonary CT angiography (523mm/s with 0.28s/rotation gantry speed). Images will be acquired using the ECG-less Cardiac software (GE Healthcare, WI, USA), without the need for patient-attached ECG leads. The system uses a wide detector coverage of 160mm to provide full heart coverage and a fast gantry speed of 0.23 seconds per rotation to perform imaging in a single cardiac cycle. An estimation of the heart rhythm must be provided, based on the heart rhythm the scanner simulates an ECG signal. This simulated ECG signal provides virtual gating of the scan. Advanced software tools including SmartPhase (automated phase selection) and SnapShot Freeze 2 (optimized volume registration) will be used. After a short delay of 5-12 sec, allowing contrast to pass from the pulmonary circulation into the aorta and coronary arteries, a coronary CT angiography will be performed using the same contrast bolus.

SUMMARY:
Chest pain represents a common reason for consultation to emergency room. This symptom can be explained by a broad spectrum of conditions, from benign musculoskeletal or esophageal pain to life-threatening disease such as aortic dissection, pulmonary embolism, and myocardial infarction.

There are already different diagnostic tools to quickly identify most dangerous diseases, for example electrocardiogram, blood samples with specific markers of cardiac injury, chest X-ray and echography. In case a doubt of disease is raised after the first clinical evaluation, it is possible to proceed with more complex, expensive and invasive examinations, namely a computed tomography (CT) scan or an invasive coronary angiography (ICA).

CT scan allows the diagnosis of various conditions such as pleural, pulmonary, pericardial and vascular disease such as pneumonia, pneumothorax, pleural and pericardial fluid, pulmonary embolism (PE), acute aortic dissection (AOD). In order to see the pulmonary, aortic and coronary arteries, a contrast injection is needed. Moreover, since the heart and the aortic root are continuously moving, specific technical measures to obtain good quality images are needed.

Recently, a new CT scan system has been developed. It allows to obtain good quality images of the heart and aortic root using an estimated heart rhythm, without ECG-gating. This allows to perform a CT scan of the heart in a reduced amount of time, and without need for controlling heart rate. Moreover, it is possible to obtain information on both aortic, coronary, and pulmonary artery with the same contrast injection. This may be of great interest in the context of patients presenting at the emergency room with chest pain and with a suspicion of pulmonary embolism, myocardial infarction, or aortic dissection, since with a single fast exam it is possible to rule out all these conditions.

Coronary arteries are very small vessels, and the accuracy of this new technique in identifying a significant obstruction is still to be proved. At present, patients with chest pain and a suspicion of myocardial infarction undergo an invasive coronary angiography. If this new tool proves to be reliable, it will be possible to reduce the number of useless invasive examination in patients in which the presence of coronary artery disease (CAD) is ruled-out. In addition, the CT scan can help quickly and effectively plan treatment when worrying abnormalities are detected in the coronary arteries that are associated with a higher risk.

Therefore, this clinical trial (further on referred to as "trial") will evaluate the investigational medicinal product (IMP), ECG-less Revolution Apex Elite system (GE Healthcare, Waukesha, WI -USA) for the diagnosis of coronary artery disease. The purpose of this trial is to learn about: the accuracy of this new CT system compared to the gold standard invasive coronary angiography in diagnosing coronary artery disease. The number of patients receiving an alternative diagnosis such as pulmonary embolism, aortic dissection, pulmonary, pleural or pericardial disease will be evaluated. Finally, the prognostic predictive value of the CT compared with ICA, in predicting myocardial infarction, coronary revascularization, and cardiac death at a follow-up of 18 months will be assessed. Patient will undergo a computer tomography examination with this new technique, evaluating both pulmonary, aortic, and coronary arteries. Then, as indicated by current guidelines, they will undergo an invasive coronary angiography.

DETAILED DESCRIPTION:
1. Study Rationale The aim is to investigate the potential role of CCTA in patients presenting to the emergency room with thoracic pain and elevated troponins. Using a single contrast bolus and a lower radiation dose, the new ECG-less CCTA could help exclude life-threatening conditions such as PE and AAD, while providing valuable information about the coronary arteries. Patients with normal coronary arteries could be safely discharged without invasive examinations, thus avoiding pro-cedural risks and optimizing both time and resources for medical institutions. However, since the diagnostic role of ECG-less CCTA in ACS has not yet been demonstrated, current guidelines and best practices will be followed in the management of enrolled patients. Decisions regard-ing PCI will be based on coronary angiography, coronary physiology, and intravascular imaging, as currently recommended by international guidelines.

   The negative and positive predictive value of the ECG-less CCTA compared to the standard of care (ICA) in patients clinically considered at risk for NSTEMI will be assessed. Additionally, the prognostic predictive value of CCTA in this clinical context, in compari-son to ICA will be evaluated. If the prognostic value of CCTA is similar to that of ICA, it will be possible to reduce the use of invasive procedures in favor of non-invasive exams, thereby saving time, contrast, and radia-tion dose for the patient.
2. Primary Objectives

   * Evaluate the diagnostic accuracy of the non-ECG-gated CCTA in diagnosing CAD compared to the gold standard (ICA) in terms of negative and positive predictive value, sensitivity, and specificity.
   * Assess the accuracy in excluding high-risk CAD such as LM, proximal LAD and multivessel disease.
   * Describe the proportion of patients diagnosed as NSTE-ACS according to the ESC guidelines who will receive an alternative diagnosis thanks to the CCTA, in particular PE and AAD.
3. Secondary Objectives

   * Assess the capacity of the non-ECG-gated CCTA in predicting the mid and long-term out-come compared to the ICA.
   * Investigate the possibility of applying the tool of FFR-CT calculation at images obtained by means of non-ECG-gated CCTA.
4. Study Design Prospective, single-center, double-blinded study.
5. Study Population Patients presenting at the ER with acute chest pain and either a diagnosis of NSTEMI at "high-risk" according to the 2023 ESC guidelines on ACS or a troponin value in the "observe pathway" and a high clinical suspicion of MI.
6. Study protocol Patients presenting with acute chest pain and elevated troponin either in the "rule-in" or "ob-serve pathway" according to ESC guidelines on ACS will be offered to participate to this study evaluating the role of non-ECG-gated CTA in patients with NSTEMI. After giving the consent, patients will be sent for non-ECG-gated CTA for the evaluation of coronary arteries, ascendent aorta and pulmonary arteries. After the CT and within 24 hours, patients will undergo ICA. Both the patient and the interventional cardiologist will be blinded to the result of the CT, the only exception being the diagnosis of a disease other than CAD which is considered responsible for the clinical presentation. The analysis of the CT images will be repeated in a core lab by the consensus of two radiologist with a wide experience in CCTA. Readers will be blinded to clini-cal data and ICA results.

ECG-less CT Patients will undergo scanning with a Revolution Apex Elite system (GE Healthcare, WI, USA), using hyperdrive pulmonary CT angiography (523mm/s with 0.28s/rotation gantry speed). Images will be acquired using the ECG-less Cardiac software (GE Healthcare, WI, USA), without the need for patient-attached ECG leads. The system uses a wide detector coverage of 160mm to provide full heart coverage and a fast gantry speed of 0.23 seconds per rotation to perform imaging in a single cardiac cycle. An estimation of the heart rhythm must be provided, which is always available since emergency patients are already monitored with finger pulse oximeter. Based on the heart rhythm the scanner simulates an ECG signal. This simulated ECG signal provides virtual gating of the scan. Acquisition can be performed over one full heart cycle, three-quarters, or half cycle, depending on heart rate. Advanced software tools including SmartPhase (automated phase selection) and SnapShot Freeze 2 (optimized volume registration) will be used to enhance image quality and correct for motion. After a short delay of 5-12 sec, allowing contrast to pass from the pulmonary circulation into the aorta and coronary arteries, a coronary CT angiography will be performed using the same contrast bolus. No additional contrast will be administered for cardiac imaging. No intravenous β-blocker or sublingual nitroglycerin will be administered. The total added exam time (including heart rhythm assessment, scan preparation, delay, and the acquisition itself) is estimated at 1-2 minutes.

Invasive coronary angiography and revascularization Patients will undergo an ICA following local and international best practices. The UZ Brussel in-terventional department is a high-volume center with experience in complex percutaneous coronary interventions (PCI). The procedures will be performed with trans-radial access when feasible. Any attention will be paid to reduce the total amount of contrast.

In case of moderate stenosis, the operator will use the invasive FFR to indicate PCI. The use of intravascular imaging is encouraged.

In case of significant CAD, patients will be treated with PCI following the ESC guidelines. The choice of interventional technique and DAPT regimen is left to the operator and the treating cardiologist.

Complete revascularization will be pursued either during the same hospitalization or within one month.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years old
* Admission at the ER with acute chest pain and at least one of the follow-ing:

  1. ECG abnormality;
  2. positive rule-in criteria according to the ESC guidelines (hs-cTnT ≥ 52 in at least one assay or 1h ∆ ≥ 5);
  3. troponine value in the "observe pathway" (hs-cTnT ≥ 12 in at least one assay or 1h ∆ ≥ 3) AND a high clinical suspicion of MI.

Exclusion Criteria:

* Indication for urgent ICA (ST-elevation, hemodynamic or electric instabil-ity, refractory chest pain, mechanical complications)
* eGFR < 30 ml/min
* Previous coronary stenting
* Previous CABG
* Recent ACS within 6 months
* Known severely reduced ejection fraction (EF < 30%)
* Contrast allergy
* Inability to provide informed consent
* Limited life expectancy < 2 years due to non-cardiac conditions
* Pregnant and breast-feeding women
* Known congenital heart disease
* Atrial fibrillation

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of ECG-less CCTA for detecting obstructive coronary artery disease (defined as luminal narrowing ≥ 50%), compared to invasive coronary angiography | Up to 12 weeks
  In both studies, sensitivity, specificity, positive and negative predictive value will be calculated. Diagnostic accuracy will be assessed using the McNemar test to compare CCTA with ICA. Cohen's Kappa agreement test will be used to evaluate agreement in diagnostic categorization between the two modalities.

SECONDARY OUTCOMES:
Accuracy of CCTA in detecting high-risk CAD such as LM, proximal LAD and multivessel disease compared to invasive coronary angigoraphy | Up to 12 weeks
  Accuracy of CCTA in detecting high-risk CAD such as LM, proximal LAD and multivessel disease compared to invasive coronary angigoraphy

OTHER OUTCOMES:
Possibility of CT-derived FFR in ECG-less CCTA | Up to 12 weeks
  We will explore the feasibility of performing fractional flow reserve (FFR)-CT analysis on ECG-less CCTA images. The added diagnostic value of FFR-CT will be evaluated comparing diagnostic accuracy of CCTA with and without FFR, using ICA as the reference.
Other conditions rather than CAD | Up to 12 weeks
  The diagnosis of conditions other than CAD such as aortic dissection, pulmonary embolism, pneumonia, pleural fluid, pneumothorax, and pericardial fluid will be recorded
Outcome prediction of ECG-less CCTA compared to ICA | at 18 months follow up
  A follow-up at 18 months will assess the occurrence of adverse events (ischemia-driven revascularization, myocardial infarction, and cardiac death). The groups of patients with positive and negative CT scan and ICA will be compared using Chi-squared test or Fisher's exact test as appropriate. For the analysis of binary outcomes, logistic regression will be utilized to establish the binary classifier for ROC curve analysis. Kaplan-Meier curves will be used to describe the event-free survival; differences between groups will be tested with the Log-Rank test. Renal function will be monitored by assessing eGFR at the time of hospitalization, before discharge, and at 18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

REFERENCES:
- [Background] Kofoed KF, Engstrom T, Sigvardsen PE, Linde JJ, Torp-Pedersen C, de Knegt M, Hansen PR, Fritz-Hansen T, Bech J, Heitmann M, Nielsen OW, Hofsten D, Kuhl JT, Raymond IE, Kristiansen OP, Svendsen IH, Dominguez Vall-Lamora MH, Kragelund C, Hove JD, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Jorgensen E, Klovgaard L, Bang LE, Helqvist S, Galatius S, Pedersen F, Abildgaard U, Clemmensen P, Saunamaki K, Holmvang L, Gislason G, Kelbaek H, Kober LV. Prognostic Value of Coronary CT Angiography in Patients With Non-ST-Segment Elevation Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Mar 2;77(8):1044-1052. doi: 10.1016/j.jacc.2020.12.037. PMID 33632478
- [Background] Linde JJ, Hove JD, Sorgaard M, Kelbaek H, Jensen GB, Kuhl JT, Hindso L, Kober L, Nielsen WB, Kofoed KF. Long-Term Clinical Impact of Coronary CT Angiography in Patients With Recent Acute-Onset Chest Pain: The Randomized Controlled CATCH Trial. JACC Cardiovasc Imaging. 2015 Dec;8(12):1404-1413. doi: 10.1016/j.jcmg.2015.07.015. Epub 2015 Nov 11. PMID 26577263
- [Background] Litt HI, Gatsonis C, Snyder B, Singh H, Miller CD, Entrikin DW, Leaming JM, Gavin LJ, Pacella CB, Hollander JE. CT angiography for safe discharge of patients with possible acute coronary syndromes. N Engl J Med. 2012 Apr 12;366(15):1393-403. doi: 10.1056/NEJMoa1201163. Epub 2012 Mar 26. PMID 22449295
- [Background] Hoffmann U, Truong QA, Schoenfeld DA, Chou ET, Woodard PK, Nagurney JT, Pope JH, Hauser TH, White CS, Weiner SG, Kalanjian S, Mullins ME, Mikati I, Peacock WF, Zakroysky P, Hayden D, Goehler A, Lee H, Gazelle GS, Wiviott SD, Fleg JL, Udelson JE; ROMICAT-II Investigators. Coronary CT angiography versus standard evaluation in acute chest pain. N Engl J Med. 2012 Jul 26;367(4):299-308. doi: 10.1056/NEJMoa1201161. PMID 22830462
- [Background] Wang K, Zhang Y, Chen B, Ren H. Comparing image quality of coronary CT angiography with and without ECG-gating in wide-detector CT. Front Cardiovasc Med. 2025 Apr 11;12:1570743. doi: 10.3389/fcvm.2025.1570743. eCollection 2025. PMID 40290191
- [Background] Linde JJ, Kelbaek H, Hansen TF, Sigvardsen PE, Torp-Pedersen C, Bech J, Heitmann M, Nielsen OW, Hofsten D, Kuhl JT, Raymond IE, Kristiansen OP, Svendsen IH, Vall-Lamora MHD, Kragelund C, de Knegt M, Hove JD, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Jorgensen E, Klovgaard L, Bang LE, Hansen PR, Helqvist S, Galatius S, Pedersen F, Abildgaard U, Clemmensen P, Saunamaki K, Holmvang L, Engstrom T, Gislason G, Kober LV, Kofoed KF. Coronary CT Angiography in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. J Am Coll Cardiol. 2020 Feb 11;75(5):453-463. doi: 10.1016/j.jacc.2019.12.012. PMID 32029126
- [Background] Meier D, Andreini D, Cosyns B, Skalidis I, Storozhenko T, Mahendiran T, Assanelli E, Sonck J, Roosens B, Rotzinger DC, Qanadli SD, Tzimas G, Muller O, De Bruyne B, Collet C, Fournier S. Usefulness of FFR-CT to exclude haemodynamically significant lesions in high-risk NSTE-ACS. EuroIntervention. 2025 Jan 6;21(1):73-81. doi: 10.4244/EIJ-D-24-00779. PMID 39468963
- [Background] Gray AJ, Roobottom C, Smith JE, Goodacre S, Oatey K, O'Brien R, Storey RF, Curzen N, Keating L, Kardos A, Felmeden D, Lee RJ, Thokala P, Lewis SC, Newby DE; RAPID-CTCA Investigators. Early computed tomography coronary angiography in patients with suspected acute coronary syndrome: randomised controlled trial. BMJ. 2021 Sep 29;374:n2106. doi: 10.1136/bmj.n2106. PMID 34588162
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Thomsen B, Nabipoor A, Asadian S, Reiser I, Cotella J, Okerlund D, Challman M, Landeras L, Chalian H. Coronary computed tomography angiography without ECG leads; A feasibility study. Curr Probl Diagn Radiol. 2025 Apr 29:S0363-0188(25)00090-8. doi: 10.1067/j.cpradiol.2025.04.019. Online ahead of print. PMID 40328582
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Background] Mancini GBJ, Leipsic J, Budoff MJ, Hague CJ, Min JK, Stevens SR, Reynolds HR, O'Brien SM, Shaw LJ, Manjunath CN, Mavromatis K, Demkow M, Lopez-Sendon JL, Chernavskiy AM, Gosselin G, Schuchlenz H, Devlin GP, Chauhan A, Bangalore S, Hochman JS, Maron DJ. CT Angiography Followed by Invasive Angiography in Patients With Moderate or Severe Ischemia-Insights From the ISCHEMIA Trial. JACC Cardiovasc Imaging. 2021 Jul;14(7):1384-1393. doi: 10.1016/j.jcmg.2020.11.012. Epub 2021 Jan 13. PMID 33454249
- [Background] Andreini D, Pontone G, Mushtaq S, Bartorelli AL, Bertella E, Antonioli L, Formenti A, Cortinovis S, Veglia F, Annoni A, Agostoni P, Montorsi P, Ballerini G, Fiorentini C, Pepi M. A long-term prognostic value of coronary CT angiography in suspected coronary artery disease. JACC Cardiovasc Imaging. 2012 Jul;5(7):690-701. doi: 10.1016/j.jcmg.2012.03.009. PMID 22789937